CLINICAL TRIAL: NCT04214847
Title: One- Year Follow up of Two Models of Ahmed Glaucoma Valves (S2 and FP7) in Refractory Glaucoma
Brief Title: The Outcome of Ahmed Glaucoma Valve in Difficult Glaucoma Cases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, khaled hamdi elbaklish, assistant professor in ophthalmology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FWA000017585 FMASU19/2017
Record Dates: First submitted 2019-12-22; First posted 2020-01-02 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Glaucoma, Open-Angle; Glaucoma Secondary; Glaucoma, Neovascular
Keywords: glaucoma-ahmed-valve-S2-FP7-IOP-encapsulation
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma, Neovascular

STUDY DESIGN:
Intervention Model Description: comparing clinical outcome variables (IOP, number of glaucoma medications, visual acuity, and complications) after using S2 and FP7 models of Ahmed Glaucoma Valves.
Who Masked: Participant, Investigator
Masking Description: Coin test to choice the participants for both groups and reduce bias. Single surgeon ,highly expert in glaucoma to minimize unnecessary postoperative result changes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- polypropylene plate of Ahmed Glaucoma Valve (Experimental): polypropylene plate of Ahmed Glaucoma Valve procedures were performed under local anesthesia except for children, general anesthesia was used. The polypropylene plate was primed and placed in the superotemporal quadrant after making fornix-based conjunctival flap. The valve plate was secured to sclera with 10-0 nylon sutures 10 mm posterior to the limbus. Before implantation, applying sponges soaked with Mitomycin- c 0.3 cc for three minutes on bare sclera at this quadrant. The tube was placed in the anterior chamber through a 23-gauge needle tract at the limbus. The tube left patent and viscoelastic substance injected into anterior chamber. A donor scleral graft was secured with interrupted 10-0 nylon sutures over the exposed portion of the tube. Conjunctiva was sutured with 10-0 nylon sutures.
  Interventions: Procedure: Ahmed Glaucoma Valve surgery
- silicone plate of Ahmed Glaucoma Valve (Active Comparator): silicone plate of Ahmed Glaucoma Valve procedures were performed under local anesthesia except for children, general anesthesia was used. The silicone plate was primed and placed in the superotemporal quadrant after making fornix-based conjunctival flap. The valve plate was secured to sclera with 10-0 nylon sutures 10 mm posterior to the limbus. Before implantation, applying sponges soaked with Mitomycin- c 0.3 cc for three minutes on bare sclera at this quadrant. The tube was placed in the anterior chamber through a 23-gauge needle tract at the limbus. The tube left patent and viscoelastic substance injected into anterior chamber. A donor scleral graft was secured with interrupted 10-0 nylon sutures over the exposed portion of the tube. Conjunctiva was sutured with 10-0 nylon sutures.
  Interventions: Procedure: Ahmed Glaucoma Valve surgery

INTERVENTIONS:
Procedure: Ahmed Glaucoma Valve surgery — The surgical procedure was identical for both implant types and was performed as described previously.9,14 All surgical procedures were performed under local anesthesia except for children, general anesthesia was used. The valve plate was primed and placed in the superotemporal quadrant after making fornix-based conjunctival flap. The valve plate was secured to sclera with 10-0 nylon sutures 10 mm posterior to the limbus. Before implantation, applying sponges soaked with Mitomycin- c 0.3 cc for three minutes on bare sclera at this quadrant. The tube was placed in the anterior chamber through a 23-gauge needle tract at the limbus. The tube left patent and viscoelastic substance injected into anterior chamber. A donor scleral graft was secured with interrupted 10-0 nylon sutures over the exposed portion of the tube. Conjunctiva was sutured with 10-0 nylon sutures.

SUMMARY:
The clinical difference (mean IOP, success rate, and complications) on using S2 and FP7 models of Ahmed Glaucoma Valve that had similar dimensions and different materials used for their construction in one year follow up was evaluated.

DETAILED DESCRIPTION:
Refractory glaucoma is a difficult subject; many glaucoma devices are tried to reduce IOP. Glaucoma devices is now an integral part of glaucoma surgery. AGV is commonly used. The investigators need to compare the efficiency and failure rate of two models of AGV. The point that is the biological reaction around capsule can affect the efficiency.

ELIGIBILITY:
Inclusion Criteria:

1. primary glaucoma patients with repeated failed trabeculectomy or other intraocular surgery.
2. patients had secondary glaucoma known to have a high failure rate with trabeculectomy such as neovascular, uveitis, post keratoplasty glaucoma or iridocorneal endothelial syndrome-associated glaucoma.

Exclusion Criteria:

1. patients lacked light perception, unwilling or unable to give informed consent, lived out of the area and were expected to be unavailable for follow-up visits,
2. patients had previous aqueous shunt implanted in the same eye, other external impediment to supero-temporal drainage device implantation.
3. patients had silicone oil, vitreous in the anterior chamber sufficient to require a vitrectomy.
4. patients had uveitis associated with a systemic condition like juvenile rheumatoid arthritis.
5. patients had nanophthalmos, Sturge-Weber syndrome or other conditions associated with elevated episcleral venous pressure.

   -

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2012-02-01 (Actual); Primary Completion 2014-03-12 (Actual); Study Completion 2014-07-15 (Actual)

PRIMARY OUTCOMES:
the postoperative mean IOP in both groups compared with the baseline IOP baseline IOP . | one-year follow up
  All measurements of the postoperative mean IOPs at 12 months were compared with the baseline IOP .

IPD SHARING:
Plan to Share IPD: No
in ophthalmology department-ophthalmic units-journal club

REFERENCES:
- [Derived] Elbaklish KH, Gomaa WA. A One-Year Follow-Up of Two Ahmed Glaucoma Valve Models (S2 and FP7) for Refractory Glaucoma: A Prospective Randomized Trial. Clin Ophthalmol. 2020 Mar 4;14:693-705. doi: 10.2147/OPTH.S224653. eCollection 2020. PMID 32184556